CLINICAL TRIAL: NCT02590458
Title: Feasibility of Short Breast MRI (SBMRI) for Screening Patients at High Risk for Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2015-0243; NCI-2015-02031 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Short Breast MRI Scan; SBMRI; Routine MRI; High risk for breast cancer; Screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Short Breast MRI (SBMRI) (Experimental): Routine scheduled MRI with contrast performed on women at high risk of developing breast cancer. One day after routine MRI, short breast MRI (SBMRI) with contrast performed. After SBMRI, participant completes a questionnaire about their comfort level and experience of the research scan.
  Interventions: Procedure: Short Breast MRI (SBMRI); Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Short Breast MRI (SBMRI) — One day after routine MRI, short breast MRI (SBMRI) with contrast performed. Scan will take about 10 minutes to complete.
  Other Names: SBMRI
Behavioral: Questionnaire — After SBMRI, participant completes a questionnaire about their comfort level and experience of the research scan. It should take about 10 minutes to complete the questionnaire.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to test if a short breast MRI scan (about 10 minutes) can be used for breast cancer screening in high risk people and to learn if it is as effective as a routine breast MRI scan (30-60 minutes).

DETAILED DESCRIPTION:
If you agree to take part in this study, you will have the short breast MRI scan (the scan for research purposes) with contrast on a different day than your scheduled routine MRI screening scan with contrast. You will have your routine scan the first day and the research scan at least 1 day after. The research scan will take about 10 minutes to complete.

After your short breast MRI scan is completed, you will complete a questionnaire about your comfort level and experience of the research scan. It should take about 10 minutes to complete the questionnaire.

This is an investigational study. The short breast MRI is considered investigational.

Up to 200 participants will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older female patients
2. BMRI indication: high risk screening per ACS guidelines
3. No contraindications to undergo MRI
4. Creatinine </=1.3 and GFR> 40
5. No requirement for sedation.

Exclusion Criteria:

1. <18 years
2. Male
3. Is pregnant (confirmed by the patient as Imaging Clinic standard of care) or nursing mother
4. Contraindication to Gd contrast agents
5. Previous documented history of moderate to severe hypersensitivity to Gd contrast agents
6. Contraindications to MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity of SBMRI for Detecting Breast Cancer in High Risk Participants | 1 day
  Radiologists blinded to patient outcome review images from each study independently and rate the possibility of breast cancer using BI-RADS score. BIRADS 0, 3,4, 5 considered positive, BIRADS 1 and 2 considered negative results for the analysis. Each reader's score for a given case assessed both independently and on a separate session, as consensus.

CONTACTS AND LOCATIONS:
Overall Officials: Marion E. Scoggins, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org